CLINICAL TRIAL: NCT01854307
Title: The Influence of Pneumoperitoneum on Minimal Invasive Cardiac Output Measurements
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low inclusion rate
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Principal Investigator, Ib Jammer, MD, Haukeland University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2012/1475/REK vest
Record Dates: First submitted 2013-05-13; First posted 2013-05-15 (Estimated); Last update posted 2016-01-25 (Estimated); Status verified 2016-01

CONDITIONS: Pneumoperitoneum
Keywords: Difference of; measurements; before and after
MeSH Terms: conditions — Pneumoperitoneum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pneumoperitoneum and SVV/PPV (Experimental)
  Interventions: Procedure: Pneumoperitoneum and SVV/PPV

INTERVENTIONS:
Procedure: Pneumoperitoneum and SVV/PPV

SUMMARY:
Perioperative goal directed fluid therapy may reduce complication rate after surgery. Minimal invasive cardiac output monitoring is a key method to guide fluid therapy. More operations are being performed by keyhole surgery (laparoscopy). For laparoscopy, the abdomen is filled with carbon dioxide. Increased pressure in the abdomen may influence minimal cardiac output monitoring, therefore minimal cardiac output monitoring is not recommended during laparoscopy. This study aims to validate minimal cardiac output monitoring during laparoscopy and therefore facilitate for goal directed fluid therapy.

ELIGIBILITY:
Inclusion Criteria:

* all patients >18 years scheduled for robot-assisted prostatectomy
* able to give informed consent

Exclusion Criteria:

* Patient with atrial fibrillation or other non-regular rhythm.
* Severe aorta/mitral stenosis
* Not able to give informed consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2013-05; Primary Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Change of stroke volume variation and pulse pressure variation during pneumoperitoneum | peroperative
  Change in PPV/SVV(LiDCO), PPV(Philips) and SVV/CO(TEE) in percent before and after pneumoperitoneum.

SECONDARY OUTCOMES:
Difference in measurements from different methods of minimal cardiac output monitoring. | peroperative
Effect of fluid bolus under pneumoperitoneum (responder vs. non-responder) | peroperative

CONTACTS AND LOCATIONS:
Locations (1):
- Haukeland University Hospital, Bergen, Norway